CLINICAL TRIAL: NCT07092254
Title: Patterns of Care and Outcomes in Locally Recurrent Inoperable or Metastatic Triple-Negative Breast Cancer in Selected Ex-US Countries
Brief Title: Patterns of Care and Outcomes in Locally Recurrent Inoperable or Metastatic Triple-Negative Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: DS1062-0007-NIS-EPI
Record Dates: First submitted 2025-07-18; First posted 2025-07-29 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Triple Negative Breast Cancer
Keywords: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced/metastatic TNBC: Adult patients who received a diagnosis of HR-negative and HER2-negative advanced/ metastatic TNBC any time from 1 January 2020 to 31 March 2024.
  Interventions: Drug: No drug

INTERVENTIONS:
Drug: No drug — No study drug will be administered in this non-interventional study.

SUMMARY:
This transnational noninterventional study aims to gather real-world evidence on locally recurrent inoperable (hereafter referred to as advanced) or metastatic TNBC (a/m TNBC) biomarker testing, treatment patterns by line of therapy, and outcomes to contextualize findings of TROPION-Breast02 and TROPION-Breast05 in selected settings outside the United States (US), including Canada, the United Kingdom (UK), France, and Spain.

DETAILED DESCRIPTION:
This study will document cancer characteristics, real-world cancer treatment patterns, clinical outcomes, and clinical events of interest in patients with locally recurrent inoperable or metastatic triple-negative breast cancer. No study or investigational drug will be administered in this non-interventional study; however, a retrospective review of medical records will be conducted.

ELIGIBILITY:
Patients meeting the following criteria will be included in the study:

* Histologically or cytologically documented diagnosis of HR-negative and HER2-negative locally recurrent inoperable TNBC (i.e., cannot be treated with curative intent) or advanced/metastatic TNBC from 1 January 2020 to 31 March 2024

  * Negative for estrogen receptor with < 1% of tumor cells positive for estrogen receptor (ER) on immunohistochemistry (IHC)
  * Negative for progesterone receptor with < 1% of tumor cells positive for progesterone receptor on IHC
  * Negative for HER2 with 0 or 1+ intensity on IHC or 2+ intensity on IHC and negative by in situ hybridization per the American Society of Clinical Oncology-College of American Pathologists (ASCO-CAP) HER2 guideline
  * The test documented closest to the diagnosis date should be used as the reference
* Aged at least 18 years upon diagnosis of advanced/metastatic TNBC
* Known vital status (alive or deceased) as of last available follow-up date documented within the medical record

Patients meeting any of the following exclusion criteria will not be eligible for the study:

* Diagnosis of other prior primary cancers or malignancies (except nonmelanoma skin cancer) unless curatively treated with no evidence of disease for at least 3 years before diagnosis of advanced/metastatic TNBC
* Ever received treatment as part of any clinical trial of an investigational product for cancer
* No available medical record entry in the 90 days before or after diagnosis of advanced/metastatic TNBC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients residing in Canada, France, Spain, and the United Kingdom who received a diagnosis of hormone receptor (HR)-negative and HER2-negative advanced/metastatic TNBC any time from 1 January 2020 to 31 March 2024.
Sampling Method: Non-Probability Sample
Enrollment: 760 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-04-08 (Estimated)

PRIMARY OUTCOMES:
Treatment sequencing before the diagnosis of advanced, metastatic TNBC (i.e., all treatments received for early TNBC if initially diagnosed with earlier-stage disease) | From date of initial diagnosis of early TNBC (if applicable) until diagnosis date of advanced, metastatic TNBC, up to approximately 15 months
  Treatment sequencing Includes broad categories for surgery, radiotherapy, adjuvant and neoadjuvant chemotherapy, immunotherapy, and start and stop dates of systemic therapy.
Treatment sequencing on or after the diagnosis date for advanced, metastatic TNBC | From date of initial diagnosis of advanced, metastatic TNBC until end of follow-up, up to approximately 15 months
  Treatment sequencing Includes broad categories for surgery, radiotherapy, adjuvant and neoadjuvant chemotherapy, immunotherapy, and start and stop dates of systemic therapy.
Real-world disease-free interval (rwDFI) | From the completion of treatment with curative intent (either date of breast tumor surgery or date of last dose of systemic therapy (whichever occurred last) and the first local or distant disease recurrence date, up to approximately 15 months
  Real-world disease-free interval (rwDFI) is assessed from the completion of treatment with curative intent (either date of primary breast tumor surgery or date of last dose of systemic anticancer therapy [not including endocrine therapy], whichever occurred last) and the first documented local or distant disease recurrence date
Clinician-defined real-world progression-free survival (rwPFS) | From the start of each line of therapy until end of follow up, up to approximately 15 months
  Clinician-defined rwPFS is assessed from the index date and from the start of each line of therapy.
Overall survival | From the start of each line of therapy until end of follow-up, up to approximately 15 months
  OS is assessed from the index date and from the start of each line of therapy.
Occurrence of clinical events of interest | From the start of each line of therapy until end of follow-up, up to approximately 15 months
  The occurrence of the following clinical events of interest will be assessed during each therapy line: Oral mucositis/stomatitis, Interstitial lung disease/pneumonitis, OSE, Diarrhea, Nausea/vomiting, Anemia, Neutropenia, Febrile neutropenia, Leukopenia, Lymphopenia, Thrombocytopenia.

CONTACTS AND LOCATIONS:
Overall Officials: Director, Study Director — Daiichi Sankyo

IPD SHARING:
Plan to Share IPD: No